CLINICAL TRIAL: NCT02042703
Title: Imaging Lens Changes in Exfoliation Syndrome Using Anterior Segment OCT
Brief Title: Imaging Lens Deposits in Exfoliation Syndrome
Status: Terminated | Type: Observational
Why Stopped: Unanticipated slow enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050919
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Exfoliation Syndrome; Primary Open Angle Glaucoma; Cataracts
MeSH Terms: conditions — Exfoliation Syndrome; Glaucoma, Open-Angle; Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- exfoliation syndrome: patients with exfoliation syndrome
  Interventions: Device: anterior segment OCT
- POAG: patients with primary open angle glaucoma (POAG)
  Interventions: Device: anterior segment OCT
- cataracts: patients with cataracts
  Interventions: Device: anterior segment OCT

INTERVENTIONS:
Device: anterior segment OCT

SUMMARY:
The purpose of this study is to use a special eye imaging technique, anterior segment optical coherence tomography (AS-OCT), to image the lens (the curved, transparent part of the eye that helps you to see clearly by directing images of light onto the back of your eye) and note any changes in exfoliation syndrome. Exfoliation syndrome is a common condition that has many ways of showing up in the eye, including the formation of deposits in the eye, shakiness of the lens that can complicate cataract surgery, and a higher chance of developing a type of glaucoma called exfoliation glaucoma. In this study we plan to collect images and measure exfoliation deposits on the lens with AS-OCT, which can take high resolution pictures of the eye without requiring contact with the eye. We will compare lens images of subjects with exfoliation syndrome to those of subjects with primary open angle glaucoma and cataracts. This type of imaging could be used in patients with known diagnosis of exfoliation syndrome to track disease progression and see how they respond to possible treatments. We also hope that with this imaging technology we can detect early changes in currently unaffected eyes, which could be useful for predicting which patients may develop the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of exfoliation syndrome, primary open angle glaucoma (POAG), or cataracts

Exclusion Criteria:

* Unable to provide or sign consent
* Pseudophakia
* Other prior intraocular surgery
* Other eye diseases other than refractive error

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Glaucoma and Comparehensive clinics at the duke Eye Center.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Amount of exfoliation deposits on the lens as measured by AS-OCT | 20 min (length of imaging)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States